CLINICAL TRIAL: NCT04040153
Title: A Pragmatic Trial of Parent-focused Prevention in Pediatric Primary Care
Brief Title: Guiding Good Choices for Health
Acronym: GGC4H
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kaiser Permanente (Other); Henry Ford Health System (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Margaret Kuklinski, Research Scientist, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SITE00000037; 4UH3AT009838 (NIH)
Record Dates: First submitted 2019-07-27; First posted 2019-07-31 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Adolescent Substance Use
Keywords: Substance; Alcohol; Tobacco; E-cigarette; Marijuana; Adolescent
MeSH Terms: conditions — Vaping; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: This is a cluster-randomized, pragmatic trial, with randomization at the pediatrician level and observation of intervention effects at the adolescent patient level. Using a constrained randomization approach, the study team will randomize 72 pediatricians, 24 in each healthcare system (36 intervention, 36 control), to either Intervention (GGC) or Control arms. Constraints (pediatrician panel size, pediatrician gender, and a pediatrician panel-level indicator of socioeconomic status) will ensure balance across intervention and control arms after randomization, reduce potential variability in effect sizes among pediatricians, and increase power. Patients and families are not aware of their pediatrician's assignment. Adolescents born between 6.1.2007 and 5.31.2009 and empaneled with the 72 pediatricians will participate in the study if their parent/legal guardian consents. GGC will be recommended to all parents/legal guardians of adolescents in the intervention arm.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guiding Good Choices (Experimental): Enrollment in the intervention, Guiding Good Choices, a substance use initiation prevention program, will be recommended by the pediatrician to parents of those adolescents empaneled with an intervention arm pediatrician
  Interventions: Behavioral: Guiding Good Choices
- Control (No Intervention): Parents of adolescents empaneled with a control arm pediatrician will not be offered Guiding Good Choices

INTERVENTIONS:
Behavioral: Guiding Good Choices — Guiding Good Choices is a 5-session group-based prevention program for parents of early adolescents. Weekly 2.5 hour sessions will be held at participants' primary care clinics and led by two trained interventionists. Through didactic material, video segments, interactive activities, and home practice, the curriculum teaches parents to understand the progression from individual and environmental risk and protective factors to substance use and problem behavior, enhances parenting behaviors and skills, teaches effective family management skills, strengthens parent-adolescent interactions and bonding, broadens opportunities for family involvement, teaches conflict reduction and anger management skills, and teaches adolescents skills to resist peer influences to engage in risky behavior. Parents who opt not to attend groups will be offered a self-guided intervention manual containing the same core content and video access, plus supportive coaching to motivate use and address questions.
  Other Names: Preparing for the Drug-Free Years
  Arms: Guiding Good Choices

SUMMARY:
This study evaluates the feasibility and effectiveness of implementing Guiding Good Choices (GGC), an anticipatory guidance curriculum for parents of early adolescents, in three large, integrated healthcare systems. By "parents," the study team is referring here and throughout this protocol to those adults who are the primary caregivers of children, irrespective of their biological relationship to the child. In prior community trials, GGC has been shown to prevent adolescent substance use (alcohol, tobacco, and marijuana), depressive symptoms, and delinquent behavior. This study offers an opportunity to test GGC effectiveness with respect to improving adolescent behavioral health outcomes when implemented at scale in pediatric primary care within a pragmatic trial.

DETAILED DESCRIPTION:
Fifty percent of all adolescents will use some form of illicit drugs before the end of high school, 20-25% will meet criteria for depression, and many others will engage in health compromising behaviors like delinquency and violence-with consequences for their long-term health. Evidence-based parenting interventions shown to prevent these behavioral health concerns could improve adolescent health trajectories if implemented widely in pediatric primary care. The American Academy of Pediatrics' Bright Futures recommends that pediatricians offer developmentally tailored anticipatory guidance to all parents to support their children's healthy development, but programs providing guidance are not offered universally.

This study tests the feasibility and effectiveness of implementing Guiding Good Choices, a universal, evidence-based anticipatory guidance curriculum for parents of early adolescents, in three large, integrated healthcare systems serving socioeconomically diverse families. This intervention reduced adolescent alcohol, tobacco and marijuana use, depression, and delinquent behavior in two previous randomized controlled trials. It also strengthened parenting practices and parent-adolescent relationship quality, both broadly protective against behavioral health concerns. Guiding Good Choices has the capacity to achieve population-level impact on adolescent health if made widely available through pediatric primary care. Parents trust pediatricians' advice regarding their children's well-being, and current research with socioeconomically diverse groups suggests that they are eager to participate in family-focused programs offered in primary care clinics.

Building on this body of research, the investigative team, in close cooperation with the NIH Healthcare Systems Research Collaboratory and healthcare systems partners, will conduct a cluster-randomized trial of Guiding Good Choices in 72 pediatric primary care practices, across three heterogeneous health care systems (HCS). Half of the pediatricians will be randomly assigned to the intervention arm, and half will serve as usual care controls. Using a workflow that is easy to adopt, implement and maintain, at each adolescent's 12-year-old well visit, primary care pediatricians will recommend that parents enroll in the intervention. Over 3,600 families are expected to be recruited into the trial prior to beginning intervention with them. Half will be recruited in year 2 and half in year 3.

The team will use the Reach, Effectiveness, Adoption, Implementation, and Maintenance, or RE-AIM, framework to test implementation outcomes and effectiveness, including hypothesized reductions in the study's primary outcome of substance use initiation, several secondary behavioral health problems (e.g., substance use frequency, mood symptoms and diagnoses, delinquency) and some exploratory outcomes (e.g., emergency department and inpatient service utilization) among adolescents in the intervention arm compared to those in the control arm. Data from an Adolescent Behavioral Health Survey and electronic healthcare records will be used to monitor outcomes up to 3 years post intervention. The feasibility and sustainability of implementing the intervention in each HCS, including health economic evaluation to understand costs in relation to value gained, will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent is empaneled with an intervention or control arm pediatrician in a participating clinic in one of the three healthcare systems (Kaiser Permanente Northern California, Kaiser Permanente Colorado, Henry Ford Health System)
* Adolescent is 12.00 - 12.99 years during intervention period (born between 6.1.2007 and 5.31.2009), which means that some adolescents may be 11 at baseline assessment

Exclusion Criteria:

* An intellectual, developmental or cognitive impairment that would prevent parent or adolescent from understanding the purpose of the study and measures, or, for those in the intervention arm, the Guiding Good Choices curriculum. For adolescents, exclusions will be operationalized by specific ICD-9/ICD-10 diagnostic codes documented in the EHR. For parents, impairment will be identified at the discretion of the pediatrician referring GGC or by study team members making study recruitment and intervention enrollment calls to parents.
* Parent's primary language is not English, as documented in the EHR or identified at study recruitment call

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3636 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adolescent substance use initiation (alcohol, cigarettes, e-cigarettes, and/or marijuana) through last follow-up | Final follow-up in year 5 of study
  Substance use initiation by the study's endpoint will be operationalized by a dichotomous indicator of ever use (yes/no) of alcohol, cigarettes, e-cigarettes, or marijuana formed from adolescent prospective self-reports about their lifetime use of these substances in each data collection wave. Substances will be assessed by separate items, e.g., "Have you ever used marijuana (by used we mean smoked, vaped, eaten, etc.)," "Have you ever used an e-cigarette or vaped ("Juul," "e-hookah," etc.)?" Lifetime use by last follow-up will be indicated by reported use of any of the substances in any wave. Lack of use will be indicated by no reported use of any of the substances in all waves.

SECONDARY OUTCOMES:
Prevalence of any past-year substance use (alcohol, cigarettes, e-cigarettes, marijuana) by adolescents at final follow-up | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  Past-year substance use at the study's endpoint will be assessed by a dichotomous indicator of past-year use (yes/no) of alcohol, cigarettes, e-cigarettes, or marijuana formed from separate items asking participants to report how many times in the past year they have used alcohol, cigarettes, e-cigarettes, and marijuana (e.g., "How many times in the past year have you used marijuana?"). Past-year use will be indicated by use of at least one of the substances at least once in the past year. No past-year use will be indicated by no reported use of any of the four substances in the past year.
Prevalence of any past-30-day substance use (alcohol, cigarettes, e-cigarettes, marijuana) by adolescents at final follow-up | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  Past-30-day substance use at the study endpoint will be assessed by a dichotomous indicator of past-30-day use (yes/no) of alcohol, cigarettes, e-cigarettes, or marijuana formed from separate items asking participants to report how many times in the past month they have used alcohol, cigarettes, e-cigarettes, and marijuana (e.g., "On how many days (if any) have you used marijuana in the past 30 days?"). Past-30-day use will be indicated by use of at least one of the substances on at least one day in the past 30 days. No past-30-day use will be indicated by no reported use of any of the four substances in the past 30 days.
Incidence of antisocial behavior among adolescents through final follow-up | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  Self-reported antisocial behavior by the study's endpoint will be assessed by a dichotomous indicator of lifetime participation in any antisocial behavior, measured by adolescent prospective reports at each wave of their participation in 7 behaviors (e.g., been suspended from school, stolen something worth more than $5, been arrested), each measured by a different item. Baseline assessment will ask participants whether they ever participated in these behaviors; subsequent assessments will ask about past-year participation. Lifetime antisocial behavior will be indicated by reported engagement in any of the 7 behaviors in any wave. Lack of antisocial behavior will be indicated by no engagement in any of the 7 behaviors in all waves.
Mean adolescent depression symptom score at final follow-up | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  Self-reports of depressive symptoms at the study endpoint will be assessed via the PHQ-9. This 9-item scale asks respondents to report on their depressive symptoms over the past 2 weeks (e.g., feeling down, depressed, irritable, or hopeless; feeling tired or having energy). Each item is scored 0=Not at all, 1=Several days, 2=More than half the days, 4=Nearly every day, yielding a total score between 0 and 36.
Mean adolescent anxiety symptom score at final follow-up | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  Self-reports of anxiety symptoms at the study endpoint will be assessed via the GAD-7, a 7-item scale that asks respondents to report on their anxiety symptoms over the past 2 weeks (e.g., feeling nervous, anxious or on edge; Trouble relaxing). Each of the 7 items is scored 0=Not at all, 1=Several days, 2=More than half the days, 4=Nearly every day, yielding a total score between 0 and 28.
Prevalence of past-year antisocial behavior among adolescents at final follow-up | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  Self-reported antisocial behavior at the study endpoint will be assessed by adolescent reports of their past-year participation in 7 behaviors (e.g., been suspended from school, stolen something worth more than $5, been arrested), each measured by a different item. Past-year antisocial behavior will be indicated by reported engagement in any of the 7 behaviors in any wave. Lack of past-year antisocial behavior will be indicated by no engagement in any of the 7 behaviors in the past year.

OTHER OUTCOMES:
Prevalence of substance use disorders among adolescents through final extraction | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  ICD-10 substance use disorder diagnoses recorded in the EHR through final data extraction. Any substance use disorder will be summarized at 12-month intervals beginning at baseline, through last extraction.
Prevalence of any psychiatric disorder (depression, anxiety, or conduct disorder) among adolescents through final extraction | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  ICD-10 depression, anxiety, and conduct disorder diagnoses recorded in the EHR through final data extraction. Any substance use disorder will be summarized at 12-month intervals beginning at baseline, through last extraction.
Prevalence of specialty substance use treatment services utilization by adolescents through final extraction | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  Specialty substance use treatment services utilization data extracted from the EHR. Any utilization will be summarized at 12-month intervals beginning at baseline, through study endpoint.
Prevalence of specialty mental health services utilization by adolescents through final extraction | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  Specialty mental health services utilization data extracted from the EHR. Any utilization will be summarized at 12-month intervals beginning at baseline, through study endpoint.
Prevalence of emergency department utilization by adolescents through final extraction | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  Automated emergency department utilization data extracted from the EHR. Any utilization will be summarized at 12-month intervals beginning at baseline, through study endpoint.
Prevalence of inpatient hospitalization utilization by adolescents through final extraction | 3-year follow-up (cohort 1), 2-year follow-up (cohort 2) assessments
  Automated inpatient hospitalization utilization data extracted from the EHR. Any utilization will be summarized at 12-month intervals beginning at baseline, through study endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret R Kuklinski, PhD, Principal Investigator — University of Washington; Richard F Catalano, PhD, Principal Investigator — University of Washington; Stacy A Sterling, DrPH, Principal Investigator — Kaiser Permanente
Locations (3):
- United States (3):
  - Kaiser Permanente Northern California, Oakland, California
  - Kaiser Permanente Colorado, Aurora, Colorado
  - Henry Ford Health System, Detroit, Michigan

REFERENCES:
- [Derived] Scheuer H, Kuklinski MR, Sterling SA, Catalano RF, Beck A, Braciszewski J, Boggs J, Hawkins JD, Loree AM, Weisner C, Carey S, Elsiss F, Morse E, Negusse R, Jessen A, Kline-Simon A, Oesterle S, Quesenberry C, Sofrygin O, Yoon T. Parent-focused prevention of adolescent health risk behavior: Study protocol for a multisite cluster-randomized trial implemented in pediatric primary care. Contemp Clin Trials. 2022 Jan;112:106621. doi: 10.1016/j.cct.2021.106621. Epub 2021 Nov 14. PMID 34785305